CLINICAL TRIAL: NCT04282525
Title: Monitoring of Cerebral Autoregulation in Pediatric ECMO (ECMOX 1)
Acronym: ECMOX1
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Istituto Giannina Gaslini (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: ECMOX1
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: ECMO; cerebral autoregulation
MeSH Terms: interventions — Extracorporeal Membrane Oxygenation; Hemodynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ECMO for hemodynamic or respiratory indication — ECMO for hemodynamic or respiratory indication

SUMMARY:
Children supported by Extra-Corporeal Membrane Oxygenation (ECMO) present a high risk of neurological complications and cerebral autoregulation (CA) impairment may be a risk factor. Our first objective is to investigate the feasibility of CA continuous monitoring during ECMO treatment. The second objective is to analyze the relationship between CA impairment and neurological outcome.

DETAILED DESCRIPTION:
Patients : All children treated by ECMO in the PICU of the Universitary hospital of Nantes, France and of IRCCS Giannina Gaslini Institute, Genoa, Italy

Measurements: A correlation coefficient between the variations of regional cerebral oxygen saturation (rScO2) as a surrogate of cerebral blood flow and the variations of arterial blood pressure (ABP) is calculated as an index of autoregulation (cerebral oxygenation index (COx), ICM+ software®). CA is monitored either on left (COxl) or both sides. A COx > 0.3 is considered as critical. Neurological outcome is assessed by the onset of an acute neurologic event (ANE) during the ECMO run.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years treated by ECMO

Exclusion Criteria:

* Lack of parental consent

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from 0 to 18 years treated by ECMO
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of continuous cerebral autoregulation monitoring | 12 hours before Extra-Corporeal Membrane Oxygenation
  Percentage of time when cerebral autoregulation metrics are available. cerebral autoregulation metrics variations under Extra-Corporeal Membrane Oxygenation
Feasibility of continuous cerebral autoregulation monitoring | During Extra-Corporeal Membrane Oxygenation
  Percentage of time when cerebral autoregulation metrics are available. cerebral autoregulation metrics variations under Extra-Corporeal Membrane Oxygenation
Feasibility of continuous cerebral autoregulation monitoring | 12 hours after Extra-Corporeal Membrane Oxygenation
  Percentage of time when cerebral autoregulation metrics are available. cerebral autoregulation metrics variations under Extra-Corporeal Membrane Oxygenation

SECONDARY OUTCOMES:
Correlation between cerebral autoregulation metrics and neurological outcome | 12 hours after Extra-Corporeal Membrane Oxygenation
  Correlation between the percentage of time spent in critical region of cerebral autoregulation and the onset of an acute neurological event (stroke and/or seizures and/or brain death) or not

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joram N, Beqiri E, Pezzato S, Moscatelli A, Robba C, Liet JM, Chenouard A, Bourgoin P, Czosnyka M, Leger PL, Smielewski P. Impact of Arterial Carbon Dioxide and Oxygen Content on Cerebral Autoregulation Monitoring Among Children Supported by ECMO. Neurocrit Care. 2021 Oct;35(2):480-490. doi: 10.1007/s12028-021-01201-8. Epub 2021 Mar 9. PMID 33686559
- [Derived] Joram N, Beqiri E, Pezzato S, Moscatelli A, Robba C, Liet JM, Chenouard A, Bourgoin P, Czosnyka M, Leger PL, Smielewski P. Continuous Monitoring of Cerebral Autoregulation in Children Supported by Extracorporeal Membrane Oxygenation: A Pilot Study. Neurocrit Care. 2021 Jun;34(3):935-945. doi: 10.1007/s12028-020-01111-1. Epub 2020 Oct 8. PMID 33029743